CLINICAL TRIAL: NCT02251470
Title: The Application of a Video-game System (Nintendo Wii®) as an Independent Exercise Program to Improve Mobility After Stroke - a Randomized Phase II Trial
Brief Title: Home-based Balance Training Using Wii Fit After Stroke: A Feasibility Study
Acronym: WiiMobil
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, André Golla, André Golla, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRM_01
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Stroke
Keywords: stroke; balance; exer-gaming; home-based exercises; Wii; postural balance; Nintendo; balance board; Wii-Fit; home; feasibility
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBE Wii (EG) (Experimental): Participants receive an introduction of using the Nintendo Wii by an individual mentoring for over 6 weeks (a total of 6 sessions á 60 minutes). During the following 6 weeks the participants perform the balance exercise program (wii-fit balances games) at home (instruction: min. 3 times a week for each 30 minutes).
  Interventions: Other: HBE Wii (EG)
- HBE Control (CG) (Active Comparator): Participants receive an introduction for conventional/traditional balance exercise by an individual mentoring for over 6 weeks (a total of 6 sessions á 60 minutes). During the following 6 weeks the participants perform the balance exercise program (exercises in standing and walking) at home (instruction: min. 3 times a week for each 30 minutes).
  Interventions: Other: HBE Control (CG)

INTERVENTIONS:
Other: HBE Wii (EG) — Wii-Fit Balance games (Soccer Heading, Ski Slalom, Table Tilt, Balance Bubble etc.)
  Arms: HBE Wii (EG)
Other: HBE Control (CG) — Simple balance exercises with own body weight (Single limb stance, stepping, side sways etc.)
  Arms: HBE Control (CG)

SUMMARY:
BACKGROUND: Virtual gaming systems offer new possibilities for home-based exercises (HBE) in rehabilitation. Pilot studies with stroke patients indicate that the application of Nintendo Wii® (WII) is practicable and can improve balance under clinical conditions. However, larger trials are necessary to verify these positive effects after discharge from the hospital.

AIM: This study aims to prepare and optimize a phase III trial which compares the effects of two HBE programs for stroke patients.

METHODS: A pilot study with randomized control design and repeated measures over three-months will be conducted. Twenty elderly stroke patients will be randomly allocated to an experimental group (EG) and a control group (CG). All participants will receive an introduction to a HBE program by an individual mentoring over 6 weeks. During the following 6 weeks the participants perform the HBE on their own. The EG will perform a balance exercise program using the WII, the CG will perform a balance exercise program without technical support.

Recruiting potential, the participants' acceptance of the intervention and economic aspects will be examined. Additionally, basic information about sensitivity of change and potential effect sizes regarding the proposed instruments to measure mobility are expected.

ELIGIBILITY:
Inclusion Criteria:

* cerebral infarction
* place of residence: Halle (Saale) and immediate surroundings
* television in household
* independent ambulatory (functional ambulation classification > 3)
* self-selected walking speed > 0,4 m/s

Exclusion Criteria:

* Strong visual impairment despite visual aid
* Deafness / verbal communication is not possible
* distinct mobility limitations due to comorbidity
* Body weight >120kg
* Epilepsy
* Cardiac pacemaker
* Acute psychiatric, disease/dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Feasibility | 12-weeks
  Recruiting potential, the participants' acceptance/satisfaction of the intervention and economic aspects

SECONDARY OUTCOMES:
Mobility | Baseline - after 6 weeks - after 12 weeks
  Berg Balance Scale, Dynamic Gait Index, Timed Up and Go (TUG) Test, Activities-Specific Balance Confidence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Mau, Prof. Dr., Study Director — Institute of Rehabilitation Medicine; André Golla, Study Chair — Institute of Rehabilitation Medicine
Locations (2):
- Germany (2):
  - Hospital "BG-Kliniken Bergmannstrost", Halle, Saxony-Anhalt
  - University Hospital Halle, Halle, Saxony-Anhalt

REFERENCES:
- [Derived] Golla A, Muller T, Wohlfarth K, Jahn P, Mattukat K, Mau W. Home-based balance training using Wii Fit: a pilot randomised controlled trial with mobile older stroke survivors. Pilot Feasibility Stud. 2018 Aug 25;4:143. doi: 10.1186/s40814-018-0334-0. eCollection 2018. PMID 30155268